CLINICAL TRIAL: NCT00135148
Title: Decrease of Libido of Post-Operative Male-Female Transsexuals and a Healthy Female Control Group
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Organon (Industry)
Other Study IDs: 2004/341
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Transsexualism
MeSH Terms: conditions — Transsexualism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Filling out a questionnaire on libido and possible partner relationship
Procedure: Sex steroid analysis

SUMMARY:
Participants fill out a questionnaire on libido and their possible partner relationship.

A blood sample is taken for sex steroid analysis.

DETAILED DESCRIPTION:
Participants fill out a questionnaire on libido and their possible partner relationship on the website http://www.onderzoek-libido.be.

A blood sample is taken for sex steroid analysis. The relation will be investigated between testosterone, free testosterone, sex hormone binding globulin, estradiol, DHEA and androstenedione and scores on relational and sexual satisfaction and sexual desire.

ELIGIBILITY:
Inclusion Criteria:

* Transsexual women with completed adaptation of the sex (all surgical procedures and hormonal treatments)
* The female control group must be 18-45 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2004-04; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guy T'Sjoen, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be